CLINICAL TRIAL: NCT02529111
Title: Integration of Three-dimensional Echocardiography and Fluoroscopy Imaging During the Percutaneous Closure of intAtrial Septal Defects in Children: CIA-3D-navigator.
Brief Title: Percutaneous Closure of Atrial Septal Defects in Children: Integration of 3D Echocardiography and Fluoroscopy Imaging.
Acronym: CIA3DNAVIGATOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/14/7415
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Atrial Septal Defects
Keywords: Atrial Septal Defects (ASD); Percutaneous closure
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): The "Echonavigator" software will be used on all patients. It will be used after the introduction of the percutaneous closure of ASD prosthesis. The image fusion on fluoroscopy will then be applied.
  Interventions: Device: "Echonavigator" software

INTERVENTIONS:
Device: "Echonavigator" software

SUMMARY:
The interventional catheterization allows the percutaneous treatment of congenital heart diseases as the atrial septal defect (ASD). The examination is guided by the X-rays with stochastic side effects worrying at the child's. The software "Echonavigator" allows to merge the ultrasound image and fluoroscopic. This innovative software facilitates the procedures and reduce the irradiation time in some adult procedures.

The aim of this study was to validate the image fusion in children.

DETAILED DESCRIPTION:
The software "Echonavigator" will be used after the introduction of the percutaneous closure of ASD prosthesis. The image fusion on fluoroscopy will then be applied and the bias between the generated ultrasound image and the X-ray view of the prosthesis will be measured. The center marker visible prosthesis ultrasound and fluoroscopy used as a reference marker.

ELIGIBILITY:
Inclusion Criteria:

* Weight higher than or equal to 20 kg
* Presence of an ostium secundum atrial septal defect diagnosed by transthoracic echocardiography and associated with a shunt from left to right evidenced by the significant dilation of the right cavities liable to a closure
* The ASD should have an anatomy allowing percutaneous closure according to international recommendations

Exclusion Criteria:

* Children with contraindication to transesophageal ultrasound according to international recommendations
* ADS with minor shunt without indication of closure
* Refusal to participate in the study expressed by parental authority

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Validity of the image fusion. | Day 1
  Through the fusion image will be measured by a fixed mark in 4 mm implications. This bias will be averaged in absolute terms and compared to zero through reference.
  The bias will be measured by two methods: one using the tool positioning an echo point of interest later merged fluoroscopy, the other using a fusion of 3D image possible with the second version.
  The method will be considered valid if the bias is not significantly different from 0 with a tolerance of 2 mm by 2 methods.

SECONDARY OUTCOMES:
Feasibility assessed by the number and percentage (calculated with the 95% confidence interval) for procedures for which the image fusion of the prosthesis of CIA has been successfully obtained will be noted. | Day1

OTHER OUTCOMES:
Safety assessed by the number and type of adverse effects associated with this technology will be noted on the day and the day after the procedure. | Day 2
Safety assessed by the heating degree of the ultrasound probe linked to the use of the software will be noted. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien HASCOET, MD, Principal Investigator — UH Toulouse
Locations (1):
- UH Toulouse, Toulouse, France

REFERENCES:
- [Background] RUBIO-ALVAREZ V, LIMON R, SONI J. [Intracardiac valvulotomy by means of a catheter]. Arch Inst Cardiol Mex. 1953 Apr;23(2):183-92. No abstract available. Undetermined Language. PMID 13066260
- [Background] Rashkind WJ, Miller WW. Creation of an atrial septal defect without thoracotomy. A palliative approach to complete transposition of the great arteries. JAMA. 1966 Jun 13;196(11):991-2. No abstract available. PMID 4160716
- [Background] Porstmann W, Wierny L, Warnke H. Closure of persistent ductus arteriosus without thoracotomy. Ger Med Mon. 1967 Jun;12(6):259-61. No abstract available. PMID 6045537
- [Background] King TD, Thompson SL, Steiner C, Mills NL. Secundum atrial septal defect. Nonoperative closure during cardiac catheterization. JAMA. 1976 Jun 7;235(23):2506-9. PMID 946659
- [Background] Van Aerschot I, Boudjemline Y. [Interventional cardiac catheterization in children]. Arch Pediatr. 2012 Jan;19(1):96-102. doi: 10.1016/j.arcped.2011.06.022. Epub 2011 Oct 29. French. PMID 22041595